CLINICAL TRIAL: NCT00358540
Title: An Open-label, Dose Ranging Study to Assess the Safety, Efficacy, and Pharmacokinetics of an Oral Thrombopoietin Receptor Agonist (Eltrombopag) Administered to Subjects Receiving Adriamycin and Ifosfamide (AI) Regimen
Brief Title: Dose Finding Study Of Oral Eltrombopag In Patients With Sarcoma Receiving Adriamycin And Ifosfamide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TRC105499; NCT00408837 (obsolete NCT alias)
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Thrombocytopaenia
Keywords: sarcoma; eltrombopag; thrombopoiesis; thrombocytopenia
MeSH Terms: conditions — Thrombocytopenia; Sarcoma | interventions — eltrombopag

ARMS (2):
- Group B (Experimental): Group B is a dose escalation phase designed to determine the optimal biological dose of eltrombopag in subjects with sarcoma who received chemotherapy treatment with Adriamycin and Ifosfamide
  Interventions: Drug: eltrombopag
- Group A (Experimental): Group A will be used for further exploration of the optimal biological dose (as initially established by completion of Group B), by using 2 different dosing schedules of eltrombopag.
  Interventions: Drug: eltrombopag

INTERVENTIONS:
Drug: eltrombopag — Dosing of sarcoma subjects with eltrombopag after treatment with Adriamycin and Ifosfamide.

SUMMARY:
The study will evaluate the safety and tolerability, optimal biologic dose, and pharmacokinetics of eltrombopag for patients with advanced sarcoma who have a low platelet count and are receiving ADRIAMYCIN and ifosfamide (AI) chemotherapy.

ELIGIBILITY:
Inclusion criteria:

* Adult subjects, 18 years or older
* Adequate liver and kidney function
* Prior history of ≥grade 2 thrombocytopenia (platelet nadir ≤ 75,000/microliters)
* Ability to ingest and retain oral medication
* Practice acceptable birth control
* Ability to understand and follow study requirements
* Life expectancy of at least 3 months

Exclusion criteria:

* History of platelet disorders, dysfunction, or a bleeding disorder
* Anti-coagulant used within 2 weeks prior to study start
* Females who are lactating or expecting
* History of thromboembolic events or drug induced thrombocytopenia
* History of central nervous system, brain and/or leptomeningeal metastases
* Prior surgery within 2 weeks or radiotherapy within 4 weeks of study start
* Pre-existing cardiac disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-06-01 (Actual); Primary Completion 2010-10-22 (Actual); Study Completion 2010-10-22 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability endpoints will consist of the evaluation of adverse events (AE), and changes from baseline in vital signs and clinical laboratory parameters | Approximately 42 weeks

SECONDARY OUTCOMES:
OBD will be determined by evaluating platelet count time course data, platelet nadirs, degree and duration of thrombocytopenia, and platelet count recovery from nadir | Approximately 18 weeks
Eltrombopag AUC(0-t) | Approximately 4 weeks
Doxorubicin and doxorubicinol PK | Approximately 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- United States (7):
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas

REFERENCES:
- [Background] Hayes S, Mudd PN Jr, Ouellet D, Johnson BM, Williams D, Gibiansky E. Population PK/PD modeling of eltrombopag in subjects with advanced solid tumors with chemotherapy-induced thrombocytopenia. Cancer Chemother Pharmacol. 2013 Jun;71(6):1507-20. doi: 10.1007/s00280-013-2150-9. Epub 2013 Apr 6. PMID 23564375
- [Derived] Chawla SP, Staddon A, Hendifar A, Messam CA, Patwardhan R, Kamel YM. Results of a phase I dose escalation study of eltrombopag in patients with advanced soft tissue sarcoma receiving doxorubicin and ifosfamide. BMC Cancer. 2013 Mar 16;13:121. doi: 10.1186/1471-2407-13-121. PMID 23497336
- See also: Results for study 105499 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/TRC105499?search=study&search_terms=105499#rs